CLINICAL TRIAL: NCT03784950
Title: Application of Behavioral Economics to Improve the Quality and Value of eConsult Specialty Reviews
Brief Title: Application of Behavioral Economics to Improve eConsult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Daniella Meeker, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-17-00077
Record Dates: First submitted 2018-12-05; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Quality of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rating tool only (Experimental): Rating eConsults from peer specialists in first phase
  Interventions: Behavioral: Rating tool
- Feedback only (Experimental): Receiving feedback from peer specialists in first phase
  Interventions: Behavioral: Feedback
- Rating Tool plus Feedback (Experimental): Both rating and feedback in second phase.
  Interventions: Behavioral: Rating tool; Behavioral: Feedback

INTERVENTIONS:
Behavioral: Rating tool — eConsult Specialty Reviewers are asked to rate the quality of other specialists' recently completed eConsult exchanges on the following four dimensions: 1) efforts to elicit additional information from PCPs, when needed; 2) medical decision making; 3) inclusion of educational content for PCPs, when appropriate; 4) perceived effect on the PCP-specialist relationship (i.e., overall tone of the eConsult exchange)
  Arms: Rating Tool plus Feedback; Rating tool only
Behavioral: Feedback — eConsult Specialty Reviewers receive confidential feedback via email on their performance (top performer vs not a top performer) as compared to colleagues in their specialty. Feedback is based on other reviewers ratings of their eConsult exchanges on the following four dimensions: 1) efforts to elicit additional information from PCPs, when needed; 2) medical decision making; 3) inclusion of educational content for PCPs, when appropriate; 4) perceived effect on the PCP-specialist relationship (i.e., overall tone of the eConsult exchange)
  Arms: Feedback only; Rating Tool plus Feedback

SUMMARY:
Using behavioral economics, the study objective is to increase the efficiency, quality, and timeliness of care for Los Angeles County (LAC) Department of Health Services (DHS) patients by nudging specialists toward more effective use of eConsult, a web-based consultation and communication portal for Primary Care Providers (PCPs) and specialists, improving access for patients in greatest need of specialty care.

DETAILED DESCRIPTION:
Historically, the Los Angeles County (LAC) Department of Health Services (DHS) Safety Net system has faced challenges in delivering specialty services that are timely, geographically equitable, and coordinated in a patient centered manner. Recently, LACDHS improved infrastructure through implementation of eConsult, a web-based consultation and communication portal for Primary Care Providers (PCPs) and specialists, improving access for patients in greatest need of specialty care. The study investigators will conduct a pragmatic randomized trial with the goal of increasing the efficiency, quality, and timeliness of care for LACDHS patients by nudging specialists toward more effective use of eConsult. If successful, these nudges may reduce the number and increase the value of face-to-face consults.

ELIGIBILITY:
Inclusion Criteria:

* LACDHS providers who are eConsult system users

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Rating - Medical Decision Making | Baseline to Post-Intervention, up to 12 months
  Peers' ratings of Medical Decision Making in Specialists' responses to PCPs
Rating - Application of Expected Practices | Baseline to Post-Intervention, up to 12 months
  Peers' ratings of Expected Practices in Specialists' responses to PCPs
Rating - Relationship Building | Baseline to Post-Intervention, up to 12 months
  Peers' ratings Relationship Building in Specialists' responses to PCPs
Rating - Expert Elicitation | Baseline to Post-Intervention, up to 12 months
  Peers' ratings of Specialists' skill in elicitation of information from PCPs
Rating - Educational Value | Baseline to Post-Intervention, up to 12 months
  Peers' ratings of Educational Value of eConsults

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Meeker, PhD, Principal Investigator — University of Southern California
Locations (1):
- Los Angeles County Department of Health Services, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnett ML, Yee HF Jr, Mehrotra A, Giboney P. Los Angeles Safety-Net Program eConsult System Was Rapidly Adopted And Decreased Wait Times To See Specialists. Health Aff (Millwood). 2017 Mar 1;36(3):492-499. doi: 10.1377/hlthaff.2016.1283. PMID 28264951
- [Background] Lee MS, Ray KN, Mehrotra A, Giboney P, Yee HF Jr, Barnett ML. Primary Care Practitioners' Perceptions of Electronic Consult Systems: A Qualitative Analysis. JAMA Intern Med. 2018 Jun 1;178(6):782-789. doi: 10.1001/jamainternmed.2018.0738. PMID 29801079
- [Derived] Behavioral Economics and eConsult Steering Committee; Meeker D, Friedberg MW, Knight TK, Doctor JN, Zein D, Cayasso-McIntosh N, Goldstein NJ, Fox CR, Linder JA, Persell SD, Dea S, Giboney P, Yee HF. Effect of Peer Benchmarking on Specialist Electronic Consult Performance in a Los Angeles Safety-Net: a Cluster Randomized Trial. J Gen Intern Med. 2022 May;37(6):1400-1407. doi: 10.1007/s11606-021-07002-1. Epub 2021 Sep 9. PMID 34505234